CLINICAL TRIAL: NCT01672970
Title: Multicenter, Post-marketing, Non-interventional, Observational Study in RA Patients Treated With Tocilizumab.
Brief Title: A Non-Interventional Study of RoActemra/Actemra in Patients With Moderate to Severe Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28212
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multi-center observational study will evaluate the use of RoActemra/Actemra (tocilizumab) in patients with rheumatoid arthritis. Eligible patients initiated on RoActemra/Actemra treatment according to the local label will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Moderate to severe rheumatoid arthritis according to the revised (1987) ACR criteria
* Patients in whom the treating physician has made the decision to commence RoActemra/Actemra treatment (in accordance with the local label); this can include patients who have received RoActemra/Actemra treatment within 8 week prior to the enrolment visit

Exclusion Criteria:

* Patients who have received RoActemra/Actemra more than 8 weeks prior to the enrolment visit
* Patients who have previously received RoActemra/Actemra in a clinical trial or for compassionate use
* Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational agent, whichever is longer) before starting treatment with RoActemra/Actemra
* History of autoimmune disease or any joint inflammatory disease other than rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis initiated on treatment with RoActemra/Actemra (tocilizumab)
Sampling Method: Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2012-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- Hungary (17):
  - Budapest
  - Debrecen
  - Eger
  - Esztergom
  - Győr
  - Gyula
  - Hévíz
  - Kecskemét
  - Kistarcsa
  - Miskolc
  - Nyíregyháza
  - Pécs
  - Szeged
  - Székesfehérvár
  - Szolnok
  - Szombathely
  - Veszprém

RESULTS

PARTICIPANT FLOW:
Groups:
- Rheumatoid Arthritis Participants: Participants with moderate to severe rheumatoid arthritis (RA), according to the American College of Rheumatology (ACR) criteria, in whom the attending physician decided to start treatment with tocilizumab (TCZ) (according to local label) at the time of recruitment or up to 8 week prior to the time of recruitment were observed for 6 months.
Period: Overall Study
Arm/Group | Rheumatoid Arthritis Participants
Started | 291
Treated | 290
Completed | 244
Not Completed | 47
Not completed — Lack of Efficacy | 12
Not completed — Adverse Event | 18
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 5
Not completed — Other | 9
Not completed — Enrolled but not treated | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) population included all participants who received at least one dose of tocilizumab and provided evaluable data.
Groups:
- Rheumatoid Arthritis Participants: Participants with moderate to severe RA, according to the ACR criteria, in whom the attending physician decided to start treatment with TCZ (according to local label) at the time of recruitment or up to 8 week prior to the time of recruitment were observed for 6 months.
Arm/Group | Rheumatoid Arthritis Participants
Number analyzed (Participants) | 290
Age, Continuous [Mean (Standard Deviation); unit: years] — Age was missing for one participant.
  years | 56.14 (12.26)
Sex/Gender, Customized [Number; unit: participants]
  Female | 261
  Male | 28
  Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants on TCZ Treatment at 6 Months After Treatment Initiation
Time Frame: 6 months
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- RA Participants: Participants with moderate to severe RA, according to the ACR criteria, in whom the attending physician decided to start treatment with TCZ (according to local label) at the time of recruitment or up to 8 week prior to the time of recruitment were observed for 6 months.
Arm/Group | RA Participants
Number analyzed (Participants) | 290
percentage of participants | 81 [76.8 to 86]

2. Secondary Outcome: Percentage of Participants With Systemic Manifestations of RA at Baseline
Description: Systemic manifestations of RA at baseline included anemia, fatigue, conventional risk factor(s) for cardiovascular disease, C-reactive protein (CRP) above upper limit of normal rheumatoid nodules, rheumatoid vasculitis, and interstitial lung disease.
Time Frame: Baseline
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 290
percentage of participants | 13.8 [10 to 18.3]

3. Secondary Outcome: Percentage of Participants Who Stopped DMARDs Prior to Start of Study and at Baseline
Description: DMARDs exposure was evaluated for all participants. "Prior DMARDs treatment" included participants, who were treated with DMARDs 8 weeks according to physician's discretion before being included in the study. "DMARDs treatment at baseline" included participants who were receiving DMARDs when they were included in the study and continued with this concomitant medication in addition to TCZ.
Time Frame: Prior to study (8 weeks) to Baseline
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 290
percentage of participants | 60.70 [54.8 to 66.3]

4. Secondary Outcome: Percentage of Participants With Reason for DMARDs Withdrawal at Baseline
Description: DMARDs exposure was evaluated for all participants. DMARDs treatment at baseline included participants, who were receiving DMARDs when they were included in the study and discontinued at baseline and not used as concomitant medication to TCZ.
Time Frame: Baseline
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 176
percentage of participants
  Lack of efficacy | 12.1
  Intolerance | 22.1
  Unspecified | 7.2
  Unknown | 19.3

5. Secondary Outcome: Number of Previous Biologic RA Treatments Received by Participants
Time Frame: Baseline
Population: FAS population
Measure: Number; unit: biologic treatments
Arm/Group | RA Participants
Number analyzed (Participants) | 290
biologic treatments
  Aceclofenac/Indometacin | 1
  Abatacept | 4
  Aceclofenac | 26
  Adalimumab | 83
  Aspirin | 1
  Azathiopirin | 16
  Betamethasone | 7
  Betamethasone/dipropionate/betamethasone sodium ph | 1
  Celecoxib | 6
  Certolizumab pegol | 63
  Chloropyramine | 1
  Chloroquine | 7
  Ciclosporin | 9
  Dexibuprofen | 1
  Diclofenac | 27
  Diclofenac/orphenadrine | 1
  Dipyrone | 1
  Etanercept | 77
  Etoricoxib | 28
  Flurbiprofen | 1
  Gold | 30
  Golimumab | 35
  Hydroxychloroquine | 95
  Ibuprofen | 1
  Indometacin | 2
  Infliximab | 66
  Ketoprofen | 1
  Leflunomide | 174
  Meloxicam | 29
  Methotrexate | 294
  Methylprednisolone | 277
  Nabumetone | 1
  Naproxen | 13
  Naproxen sodium | 3
  Niflumic acid | 1
  Nimesulide | 13
  Paracetamol | 6
  Paracetamol/Tramadol | 1
  Penicillamine | 1
  Penicillin G sodium | 1
  Phenylbutazone | 1
  Piroxicam | 3
  Prednisolone | 10
  Rituximab | 17
  Sulfasalazine | 171
  Tocilizumab | 2
  Tramadol | 30
  Triamcinolone | 2
  Triamcinolone acetonide | 3
  Triamcinolone hexacetonide | 1
  Valdecoxib | 1

6. Secondary Outcome: Percentage of Participants With Duration of Previous Biologic RA Treatments
Description: The duration of previous biologic RA treatments was classified in to two categories: less than (<) 6 months and greater than (>) 6 months.
Time Frame: Baseline
Population: Per protocol population included all participants who had a valid tocilizumab administration assessment at 6-month time window and without any protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 232
percentage of participants
  <6 months | 0.0
  >6 months | 100.0

7. Secondary Outcome: Percentage of Participants With Reasons for Termination of Previous Biologic RA Treatments
Description: Lack of efficacy was determined as per physicians' discretion. Intolerance was defined as the participant could not be treated due to safety reason (adverse events).
Time Frame: Baseline
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 170
percentage of participants
  Lack of efficacy | 42.1
  Intolerance | 11.7
  Unspecified | 4.5
  Unknown | 0.3

8. Secondary Outcome: Number of Participants With Reasons for Dose Modification for TCZ
Description: Only those participants that had dose modifications were reported.
Time Frame: 6 months
Population: FAS population
Measure: Number; unit: participants
Arm/Group | RA Participants
Number analyzed (Participants) | 290
participants
  Adverse event | 17
  Normalization of absolute neutrophil count | 3
  Unspecified | 6

9. Secondary Outcome: Mean Dose of TCZ at 6 Months
Description: TCZ was administered every 4 weeks according to the label. Due to the observational nature of the study, the suggested schedule was subject to changes according to physician and participant considerations.
Time Frame: 6 months
Population: FAS population. Here number of participants analyzed = participants available for the analysis of this outcome measure.
Measure: Mean (Standard Deviation); unit: milligrams per kilogram {mg/kg)
Arm/Group | RA Participants
Number analyzed (Participants) | 237
milligrams per kilogram {mg/kg) | 7.8926 (0.57949)

10. Secondary Outcome: Mean Dosing Interval of Treatment at 6 Months
Description: as for outcome 9
Time Frame: 6 months
Population: FAS population. Here number of participants analyzed = participants available for the analysis of this outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | RA Participants
Number analyzed (Participants) | 284
days | 31.79 (5.81)

11. Secondary Outcome: Percentage of Participants Discontinued From Tocilizumab for Safety And Efficacy Reasons
Description: The safety variable measured the number of participants who discontinued TCZ due to adverse reactions to TCZ, and the efficacy variable measured the participants who discontinued from TCZ due to lack of efficacy according to criteria of the treating physician.
Time Frame: 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 46
percentage of participants
  Intolerable adverse events | 6.2
  Lack of efficacy | 4.1
  Other Unspecified reason | 5.5

12. Secondary Outcome: Number of Participants With Restoration of Initial Dosing Regimen of TCZ
Description: The number of participants who reported restoration of initial dosing regimen of TCZ for 84.00, 133.00, 158.00, 2.3.00 and 206.00 days, were reported.
Time Frame: 6 months
Population: Per protocol population
Measure: Number; unit: participants
Arm/Group | RA Participants
Number analyzed (Participants) | 232
participants
  84.00 days | 1
  133.00 days | 1
  158.00 days | 2
  203.00 days | 1
  206.00 days | 1

13. Secondary Outcome: Percentage of Participants Adhered to the Dosing Regimen Recommended by Physician for TCZ
Description: A participant's adherence was calculated based on the adverse event or laboratory abnormality experienced by the participants who required dose modifications as per local TCZ label or protocol.
Time Frame: 6 months
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 290
percentage of participants
  Adverse events | 1.38
  Other reasons | 1.38

14. Secondary Outcome: Percentage of Participants on Tocilizumab Monotherapy
Description: as for outcome 9
Time Frame: 6 months
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 290
percentage of participants | 40.0 [34.3 to 45.9]

15. Secondary Outcome: Percentage of Participants With Reason for DMARD Withdrawal
Description: Objective intolerance was determined by medical observation; subjective intolerance was determined by the participant; lack of efficacy was determined by physician discretion.
Time Frame: 6 months
Population: FAS population. Here number of participants analyzed = participants available for the analysis of this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 73
percentage of participants
  Lack of efficacy | 12.3
  Intolerance | 67.1
  Oher unspecified reason | 20.5
  Withdrew informed consent | 0.7
  Other | 3.1

16. Secondary Outcome: Change From Baseline in Tender Joint Count (28 Joints) at Months 3 and 6
Description: The number of tender joints was recorded on the joint assessment form, no tenderness = 0, tenderness = 1, for 28 joints and joints were classified as tender/not tender giving a total possible tender joint count score of 0 to 28.
Time Frame: Baseline, 3 and 6 months
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure. Here "n"= participants who were evaluable for each category.
Measure: Mean (Standard Deviation); unit: joint count
Arm/Group | RA Participants
Number analyzed (Participants) | 259
joint count
  Month 3 (n=259) | -10.2703 (7.41544)
  Month 6 (n=215) | -10.6744 (7.64432)
Statistical Analysis 1: Comparison: RA Participants; Statistical analysis at Month 3; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: RA Participants; Statistical Analysis at Month 6; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Rank Test

17. Secondary Outcome: Change From Baseline in Tender Joint Count (68 Joints) at Months 3 and 6
Description: The number of tender joints was recorded on the joint assessment form, no tenderness = 0, tenderness = 1, for 68 joints and joints were classified as tender/not tender giving a total possible tender joint count score of 0 to 68.
Time Frame: Baseline, 3 and 6 months
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: joint count
Arm/Group | RA Participants
Number analyzed (Participants) | 23
joint count
  Month 3 (n=23) | -48.2904 (49.94400)
  Month 6 (n=21) | -60.0820 (51.74519)
Statistical Analysis 1: Comparison: RA Participants; Statistical Analysis at Month 3; Test type: Superiority or Other; p = 0.001, Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: RA Participants; Statistical Analysis at Month 6; Test type: Superiority or Other; p = 0.005, Wilcoxon Signed Rank Test

18. Secondary Outcome: Change From Baseline in Swollen Joint Count (28 Joints) at Months 3 and 6
Description: The number of swollen joints was recorded on the joint assessment form, no swelling = 0, swelling =1, for 28 joints and were classified as swollen/not swollen giving a total possible swollen joint count score of 0 to 28.
Time Frame: Baseline, 3 and 6 months
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: joint count
Arm/Group | RA Participants
Number analyzed (Participants) | 259
joint count
  Month 3 (n=259) | -6.6641 (6.22130)
  Month 6 (n=215) | -7.0651 (6.28047)
Statistical Analysis 1: Comparison: RA Participants; Statistical Analysis at Month 3; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: RA Participants; Statistical Analysis at Month 6; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Rank Test

19. Secondary Outcome: Change From Baseline in Swollen Joint Count (66 Joints) at Months 3 and 6
Description: The number of swollen joints was recorded on the joint assessment form, no swelling = 0, swelling =1, for 66 joints and were classified as swollen/not swollen giving a total possible swollen joint count score of 0 to 66.
Time Frame: Baseline, 3 and 6 months
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: joint count
Arm/Group | RA Participants
Number analyzed (Participants) | 20
joint count
  Month 3 (n=20) | -70.6711 (35.24487)
  Month 6 (n=17) | -80.9244 (27.34339)
Statistical Analysis 1: Comparison: RA Participants; Statistical Analysis at Month 3; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: RA Participants; Test type: Superiority or Other; p = 0.001, Wilcoxon Signed Rank Test

20. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28 Joint Count (DAS28) at Months 3 and 6
Description: DAS28 was calculated from SJC and TJC using 28 joints count, erythrocyte sedimentation rate (ESR) (millimeter per hour [mm/hr]), and Participant's Global Assessment (PGH) of disease activity (measured on a 0 to 100 mm Visual Analogue Scale (VAS) where 0=no disease activity and 100=worst disease activity). DAS28 was calculated using following formula: DAS28 = 0.56*square root (sqrt) (TJC28) + 0.28*sqrt(SJC28) + 0.70*natural logarithm (ln) (ESR) + 0.014*PGH of disease activity. Total score range: 0-10, higher score=more disease activity. DAS28 <3.2 implied low disease activity, DAS >3.2 to 5.1 implied moderate disease activity and DAS >5.1 implied high disease activity, and DAS28 <2.6 = clinical remission.
Time Frame: Baseline, 3 and 6 months
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA Participants
Number analyzed (Participants) | 250
units on a scale
  Month 3 (n=250) | 2.6156 (1.23416)
  Month 6 (n=209) | 2.2703 (1.09059)

21. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Response
Description: Clinical response assessed as per EULAR categorical DAS28 response criteria was defined as clinically meaningful improvement at a particular time point. EULAR response was based on change from baseline (CFB) in the DAS28 score and also on the actual DAS28 score at the time point so was more reflective of the current status of the participant. The DAS28 score was a measure of the participant's disease activity, based on the TJC (28 joints), SJC (28 joints), PGH (mm), and ESR (mm/hr). DAS28 total scores ranged from 0 to approximately 10. Scores <2.6 = best disease control and scores >5.1 = worse disease control. A negative CFB indicated clinically meaningful improvement. EULAR Good response: DAS28 <=3.2 and a CFB <-1.2. EULAR Moderate response: DAS28 >3.2 to ≤ 5.1 or a CFB < -0.6 to ≥ -1.2. EULAR No response: DAS28 ≤3.2 or CFB greater than or equal to (>=) -0.6, DAS28 >3.2 to <=5.1 or CFB >=-0.6 and DAS28 >5.1 or CFB >=-0.6.
Time Frame: Visit 2 (Month 1), Visit 3 (Month 2), Visit 4 (Month 3), Visit 5 (Month 4), Visit 6 (Month 5), Visit 7 (Months 6) and Visit 8 (Final Visit; within 2 weeks after 6months observation period)
Population: FAS population. Here, number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 252
percentage of participants
  Visit 2 (Month 1) | 75.2 [69.8 to 80.0]
  Visit 3 (Month 2) | 7.2 [4.5 to 10.9]
  Visit 4 (Month 3) | 3.1 [1.4 to 5.8]
  Visit 5 (Month 4) | 0.7 [0.1 to 2.5]
  Visit 6 (Month 5) | 0.3 [0.0 to 1.9]
  Visit 7 (Month 6) | 0.3 [0.0 to 1.9]
  Visit 8 (Final Visit) | 0 [0.0 to 1.3]

22. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) Score at Months 3 and 6
Description: The SDAI was a combined index for measuring disease activity in RA which reflected the numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, PGH and physician's global assessment (PhGH) of disease activity, assessed on 0-100 mm VAS where 0 = no disease activity and 100 = worst disease activity, and C-reactive protein (CRP) (milligrams per deciliter [mg/dL]). SDAI total score = 0-86. A SDAI score of <=3.3 represented clinical remission, a score of >3.4 to <=11.0 represented low disease activity, a score of >11 to <=26.0 represented moderate disease activity and a score of >26.0 represented high (or severe) disease.
Time Frame: Baseline, 3 and 6 months
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA Participants
Number analyzed (Participants) | 185
units on a scale
  Month 3 (n=185) | -45.4383 (38.24144)
  Month 6 (n=148) | -47.5846 (33.88556)
Statistical Analysis 1: Comparison: RA Participants; Statistical Analysis at Month 3; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: RA Participants; Statistical Analysis at Month 6; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Ranks Test

23. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Score at Months 3 and 6
Description: The CDAI was a combined index for measuring disease activity in RA and used to evaluate disease activity in the absence of laboratory testing of CRP and ESR. It was the numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PGH and PhGH (assessed on 0-100 mm VAS); VAS (0 = no disease activity and 100 = worst disease activity). CDAI total score = 0-76. A CDAI score of <=2.8 represented clinical remission, a score of >2.8 to <=10.0 represented low disease activity, a score of >10.0 to <=22.0 represented moderate disease activity and a score of >22.0 represented high (or severe) disease.
Time Frame: Baseline, 3 and 6 months
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA Participants
Number analyzed (Participants) | 206
units on a scale
  Month 3 (n=206) | -24.6068 (14.41937)
  Month 6 (n=173) | -26.0046 (14.58529)
Statistical Analysis 1: Comparison: RA Participants; Statistical Analysis at Month 3; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: RA Participants; Statistical Analysis at Month 6; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Ranks Test

24. Secondary Outcome: Percentage of Participants Who Achieved 20 Percent (%) Improvement in ACR (ACR20) Response
Description: ACR response was calculated based on total joint count evaluation (28 or 66/68 joint count) and other clinical and laboratory assessments. A positive ACR20 response required at least a 20% improvement (reduction) compared to baseline in swollen joint count (66 joints) and tender joint count (68 joints) and at least 3 of the following 5 assessments: participant's global assessment of pain, PGH, PhGH (all 3 assessed at 0 [good] to 100 mm [worst] VAS scale), participant assessment of disability measured by the Health Assessment Questionnaire-Disability Index (HAQ-DI) (assessed on a 0 to 3 scale, where higher scores represented higher disease activity), Acute phase reactant (CRP or ESR). A reduction in the level of and acute phase reactants was considered an improvement.
Time Frame: Baseline, 3 and 6 months
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 290
percentage of participants
  Month 3 | 3.80 [1.9 to 6.7]
  Month 6 | 4.5 [2.4 to 7.5]

25. Secondary Outcome: Percentage of Participants Who Achieved 50% Improvement in ACR (ACR50) Response
Description: ACR response was calculated based on total joint count evaluation (28 or 66/68 joint count) and other clinical and laboratory assessments. A positive ACR50 response required at least a 50% improvement (reduction) compared to baseline in swollen joint count (66 joints) and tender joint count (68 joints) and at least 3 of the following 5 assessments: (participant's global assessment of pain, PGH, PhGH (all 3 assessed at 0 [good] to 100 mm [worst] VAS scale), participant assessment of disability measured by the Health Assessment Questionnaire-Disability Index (HAQ-DI) (assessed on a 0 to 3 scale, where higher scores represented higher disease activity), and acute phase reactant (CRP or ESR). A reduction in the level of acute phase reactants was considered an improvement.
Time Frame: Baseline, 3 and 6 months
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 290
percentage of participants
  Month 3 | 3.10 [1.4 to 5.8]
  Month 6 | 1.70 [0.6 to 4.0]

26. Secondary Outcome: Percentage of Participants Who Achieved 70% Improvement in ACR (ACR70) Response
Description: ACR response was calculated based on total joint count evaluation (28 or 66/68 joint count) and other clinical and laboratory assessments. A positive ACR70 response required at least a 70% improvement (reduction) compared to baseline in swollen joint count (66 joints) and tender joint count (68 joints) and at least 3 of the following 5 assessments: (participant's global assessment of pain, PGH, PhGH (all 3 assessed at 0 [good] to 100 mm [worst] VAS scale), participant assessment of disability measured by the Health Assessment Questionnaire-Disability Index (HAQ-DI) (assessed on a 0 to 3 scale, where higher scores represented higher disease activity), and acute phase reactant (CRP or ESR). A reduction in the level of acute phase reactants was considered an improvement.
Time Frame: Baseline, 3 and 6 months
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 290
percentage of participants
  Month 3 | 1.40 [0.4 to 3.5]
  Month 6 | 1.40 [0.4 to 3.5]

27. Secondary Outcome: Percentage of Participants Who Achieved 90% Improvement in ACR (ACR90) Response
Description: ACR response was calculated based on total joint count evaluation (28 or 66/68 joint count) and other clinical and laboratory assessments. A positive ACR90 response required at least a 90% improvement (reduction) compared to baseline in swollen joint count (66 joints) and tender joint count (68 joints) and at least 3 of the following 5 assessments: (participant's global assessment of pain, PGH, PhGH (all 3 assessed at 0 [good] to 100 mm [worst] VAS scale), participant assessment of disability measured by the Health Assessment Questionnaire-Disability Index (HAQ-DI) (assessed on a 0 to 3 scale, where higher scores represented higher disease activity), and acute phase reactant (CRP or ESR). A reduction in the level of acute phase reactants was considered an improvement.
Time Frame: Baseline, 3 and 6 months
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RA Participants
Number analyzed (Participants) | 290
percentage of participants
  Month 3 | 0.70 [0.1 to 2.5]
  Month 6 | 0.70 [0.1 to 2.5]

28. Secondary Outcome: Change From Baseline in Physician Global Assessment of Disease Activity at Months 3 and 6
Description: The physician's global assessment of disease activity was assessed using a 0 to 100 mm horizontal VAS by the physician. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative change from Baseline indicated improvement.
Time Frame: Baseline, 3 and 6 months
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA Participants
Number analyzed (Participants) | 214
units on a scale
  Month 3 (n=214) | -37.3832 (21.41701)
  Month 6 (n=177) | -43.9096 (20.78387)
Statistical Analysis 1: Comparison: RA Participants; Statistical Analysis at Month 3; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: RA Participants; Statistical Analysis at Month 6; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Ranks Test

29. Secondary Outcome: Change From Baseline in Participant Global Assessment of Disease Activity at Months 3 and 6
Description: The Participant's Global Assessment of Disease Activity was assessed using a 0 to 100 mm horizontal VAS by the participant. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative change from Baseline indicated improvement.
Time Frame: Baseline, 3 and 6 months
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA Participants
Number analyzed (Participants) | 238
units on a scale
  Month 3 (n=238) | -33.2437 (24.64703)
  Month 6 (n=201) | -39.3930 (25.06551)
Statistical Analysis 1: Comparison: RA Participants; Statistical Analysis at Month 3; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: RA Participants; Statistical Analysis at Month 6; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Ranks Test

30. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Months 3 and 6
Description: The HAQ-DI was a participant self-reported questionnaire for assessing the extent of a participant's functional ability. It consisted of 20 questions in 8 categories (dressing and grooming, rising, eating, walking, reach, grip, hygiene, and carrying out daily activities). Each question had 4 response options, ranging from 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. The HAQ-DI scale was an average of all the scores and ranged from 0 to 3, where higher scores represented higher disease activity.
Time Frame: Baseline, 3 and 6 months
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA Participants
Number analyzed (Participants) | 205
units on a scale
  Month 3 (n=205) | 0.4766 (0.62768)
  Month 6 (n=173) | 0.5497 (0.63257)
Statistical Analysis 1: Comparison: RA Participants; Statistical Analysis at Month 3; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Ranks Test
Statistical Analysis 2: Comparison: RA Participants; Statistical Analysis at Month 6; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Ranks Test

31. Secondary Outcome: Change From Baseline in Participant's Assessment of Fatigue Using VAS at Months 3 and 6
Description: Fatigue was evaluated by a VAS. Participants marked on a 100 mm horizontal VAS the level of fatigue that they have experienced, ranging from 0 (no fatigue) to 100 (extreme fatigue).
Time Frame: Baseline, 3 and 6 months
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA Participants
Number analyzed (Participants) | 198
units on a scale
  Month 3 (n=198) | -26.4192 (26.05482)
  Month 6 (n=162) | -32.5000 (25.94984)
Statistical Analysis 1: Comparison: RA Participants; Statistical Analysis at Month 3; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: RA Participants; Statistical Analysis at Month 6; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Rank Test

32. Secondary Outcome: Change From Baseline in Participant's Assessment of RA-Related Pain Using VAS at Months 3 and 6
Description: Severity of pain was evaluated by a VAS. Participants marked on a 100 mm horizontal VAS the severity of pain that they had experienced because of their RA, ranging from 0 (no pain) to 100 (unbearable pain).
Time Frame: Baseline, 3 and 6 months
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA Participants
Number analyzed (Participants) | 239
units on a scale
  Month 3 (n=239) | -31.0586 (23.45828)
  Month 6 (n=194) | -36.9948 (25.95782)
Statistical Analysis 1: Comparison: RA Participants; Statistical Analysis at Month 3; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: RA Participants; Statistical Analysis at Month 6; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Rank Test

33. Secondary Outcome: Change From Baseline in Particpant's Assessment of RA Morning Stiffness Assessed Using VAS at Months 3 and 6
Description: Morning stiffness was defined by the time elapsed between the time of usual awakening (even if not in the morning) and the time the participant was as limber as he/she would be during a day involving typical activities. Morning stiffness was assessed on a 100 mm VAS, where 0= none and 100= very severe.
Time Frame: Baseline, 3 and 6 months
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA Participants
Number analyzed (Participants) | 151
units on a scale
  Month 3 (n=151) | -25.7285 (26.61877)
  Month 6 (n=117) | -32.5043 (26.08792)
Statistical Analysis 1: Comparison: RA Participants; Statistical Analysis at Month 3; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: RA Participants; Statistical Analysis at Month 6; Test type: Superiority or Other; p = 0.000, Wilcoxon Signed Rank Test

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: FAS population
Arm/Group | Rheumatoid Arthritis Participants
Serious Adverse Events (participants affected / at risk) | 17/290
Other Adverse Events (participants affected / at risk) | 108/290
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rheumatoid Arthritis Participants (N=290)
Leucocytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 2
Vertigo (Ear and labyrinth disorders) | 1
Keratitis (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Ulcerative keratitis (Eye disorders) | 1
Corneal disorders (Eye disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 2
Glomerular filtration rate increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 2
Neutrophil count increase (Investigations) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypotonia (Nervous system disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
Embolism (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rheumatoid Arthritis Participants (N=290)
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 5
Granulocytopenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Extrasystoles (Cardiac disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Chest pain (General disorders) | 1
Drug ineffective (General disorders) | 2
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Hepatobiliary disease (Hepatobiliary disorders) | 1
Acarodermatitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 4
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 2
Erysipelas (Infections and infestations) | 2
Fungal skin infection (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Influenza (Infections and infestations) | 9
Oral herpes (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 5
Blood cholesterol increased (Investigations) | 1
Blood pressure increased (Investigations) | 9
Blood triglycerides increased (Investigations) | 1
Gamma-glutamyl transferase increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 5
Liver function test abnormal (Investigations) | 1
Lymphocyte count increased (Investigations) | 1
Mycobacterium tuberculosis complex test positive (Investigations) | 1
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 1
Transaminases increased (Investigations) | 3
Weight decreased (Investigations) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Cervicobrachial syndrome (Nervous system disorders) | 1
Hypotonia (Nervous system disorders) | 1
Trigeminal neuralgia (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2
Cholecystectomy (Surgical and medical procedures) | 1
Tooth extraction (Surgical and medical procedures) | 3
Hypertension (Vascular disorders) | 5
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.